CLINICAL TRIAL: NCT04347200
Title: Registry Dedicated to Assess the Risk of Ischemic and Hemorrhagic Complications of Long-term Antithrombotic Therapy in Patients With Chronic Coronary Syndromes
Brief Title: REGistry of Long-term AnTithrombotic TherApy-1
Acronym: REGATTA-1
Status: Recruiting | Type: Observational
Sponsor: National Medical Research Center for Cardiology, Ministry of Health of Russian Federation (Other Government)
Responsible Party: Sponsor
Other Study IDs: REGATTA119021970
Record Dates: First submitted 2020-04-10; First posted 2020-04-15 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Coronary Artery Disease (CAD) (E.G., Angina, Myocardial Infarction, and Atherosclerotic Heart Disease (ASHD)); Peripheral Artery Disease
Keywords: Coronary Artery Disease, Peripheral Artery Disease
MeSH Terms: conditions — Coronary Artery Disease; Angina Pectoris; Myocardial Infarction; Peripheral Arterial Disease | interventions — Platelet Aggregation Inhibitors; Anticoagulants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — whole blood, serum, white cells, urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Antiplatelet Drug — single or dual antiplatelets, triple antithrombotic therapy
  Other Names: anticoagulant Drug

SUMMARY:
To assess the rates of ischemic and hemorrhagic complications of long-term antithrombotic therapy in patients with chronic coronary syndromes

DETAILED DESCRIPTION:
The register is a Russian prospective single-center observational study of patients who have indications for long-term antithrombotic therapy in connection with chronic coronary syndromes

ELIGIBILITY:
Inclusion Criteria:

* coronary artery disease , confirmed by history of myocardial infarction, or revascularization, or definitive evidence of CAD on imaging

Exclusion Criteria:

* Subjects who are unwilling or unable to provide informed consent.
* Acute coronary syndrome within 12 months before inclusion
* Severe chronic heart failure (NYHA IV)
* Stroke within 6 months before inclusion
* Severe liver or muscle disease
* Severe kidney disease / renal failure with creatinine > 3 mg/dl
* Conceivable impossibility to come in touch with the patient or his family at 1-year after the intervention -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized or outpatients with confirmed chronic coronary syndromes
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2015-01-15 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
composite of major adverse cardiovascular events (MACE) | inclusion up to 5 years
  stroke, myocardial infarction, stent thrombosis [definite or probable], or urgent revascularization, cardiac death
composite of any bleeding events | inclusion up to 5 years
  major, clinically relevant nonmajor, minor (BARC, ISTH)

SECONDARY OUTCOMES:
Severity of peripheral atherosclerosis | inclusion
  Assessment will be performed with the use of duplex scanning
Mutations in following genes | inclusion
  CYP2C19*, ABCB1

CONTACTS AND LOCATIONS:
Overall Officials: Elizaveta Panchenko, PhD, Principal Investigator — National Medical Research Center for Cardiology, Ministry of Health of Russian Federation
Locations (1):
- National Medical Research Center for Cardiology, Ministry of Health of Russian Federation, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No
Individual participant data that underlie the results reported in the article after deidentification (text, tables, figures)

REFERENCES:
- [Background] Komarov AL, Shakhmatova OO, Korobkova VV. [The balance of benefit and risk in prescribing antithrombotic therapy for patients with coronary artery disease. How to deal with the gastrointestinal bleeding problem?]. Kardiologiia. 2020 Aug 11;60(7):115-124. doi: 10.18087/cardio.2020.7.n1159. Russian. PMID 33155950
- [Background] Shakhmatova OO, Komarov AL, Krivosheeva EN, Dobrovolsky AB, Titaeva EV, Amelyushkina VA, Gomyranova NV, Panchenko EP. [Albuminuria as a marker of atherosclerosis burden and a possible predictor of adverse events in patients with polyvascular disease]. Ter Arkh. 2023 Nov 3;95(9):763-768. doi: 10.26442/00403660.2023.09.202434. Russian. PMID 38158919
- [Background] Eikelboom JW, Connolly SJ, Bosch J, Dagenais GR, Hart RG, Shestakovska O, Diaz R, Alings M, Lonn EM, Anand SS, Widimsky P, Hori M, Avezum A, Piegas LS, Branch KRH, Probstfield J, Bhatt DL, Zhu J, Liang Y, Maggioni AP, Lopez-Jaramillo P, O'Donnell M, Kakkar AK, Fox KAA, Parkhomenko AN, Ertl G, Stork S, Keltai M, Ryden L, Pogosova N, Dans AL, Lanas F, Commerford PJ, Torp-Pedersen C, Guzik TJ, Verhamme PB, Vinereanu D, Kim JH, Tonkin AM, Lewis BS, Felix C, Yusoff K, Steg PG, Metsarinne KP, Cook Bruns N, Misselwitz F, Chen E, Leong D, Yusuf S; COMPASS Investigators. Rivaroxaban with or without Aspirin in Stable Cardiovascular Disease. N Engl J Med. 2017 Oct 5;377(14):1319-1330. doi: 10.1056/NEJMoa1709118. Epub 2017 Aug 27. PMID 28844192
- [Background] Darmon A, Sorbets E, Ducrocq G, Elbez Y, Abtan J, Popovic B, Ohman EM, Rother J, Wilson PF, Montalescot G, Zeymer U, Bhatt DL, Steg PG; REACH Registry Investigators. Association of Multiple Enrichment Criteria With Ischemic and Bleeding Risks Among COMPASS-Eligible Patients. J Am Coll Cardiol. 2019 Jul 2;73(25):3281-3291. doi: 10.1016/j.jacc.2019.04.046. PMID 31248549
- [Background] Komarov A, Panchenko E, Dobrovolsky A, Karpov Y, Deev A, Titaeva E, Davletov K, Eshkeeva A, Markova L. D-dimer and platelet aggregability are related to thrombotic events in patients with peripheral arterial occlusive disease. Eur Heart J. 2002 Aug;23(16):1309-16. doi: 10.1053/euhj.2001.3116. PMID 12175668
- [Background] Komarov AL, Shakhmatova OO, Muraseeva VG, Novikova ES, Guskova EV, Panchenko EP. Proton pump inhibitors receiving and prognosis of patients after scheduled percutaneous coronary interventions. Ter Arkh. 2018 Sep 20;90(9):92-100. doi: 10.26442/terarkh201890992-100. PMID 30701742
- [Background] Darmon A, Bhatt DL, Elbez Y, Aboyans V, Anand S, Bosch J, Branch KR, Connolly SJ, Dyal L, Eikelboom JW, Fox KAA, Keltai K, Probstfield J, Yusuf S, Abtan J, Sorbets E, Eagle KA, Ducrocq G, Steg PG. External applicability of the COMPASS trial: an analysis of the reduction of atherothrombosis for continued health (REACH) registry. Eur Heart J. 2018 Mar 1;39(9):750-757a. doi: 10.1093/eurheartj/ehx658. PMID 29186454
- [Background] Komarov AL, Shahmatova OO, Korobkova VV, Kurilina EV, Shuleshova AG, Panchenko EP. [Gastric mucosa condition in patients with coronary artery disease and high risk of gastrointestinal bleeding (register REGATTA-1)]. Ter Arkh. 2021 Dec 15;93(12):1457-1462. doi: 10.26442/00403660.2021.12.201224. Russian. PMID 36286673
- [Background] Shakhmatova OO, Komarov AL, Korobkova VV, Yarovaya EB, Andreevskaya MV, Shuleshova AG, Panchenko EP. [Upper gastrointestinal bleeding in patients with stable coronary artery disease (registry of antithrombotic therapy "REGATcapital TE, CyrillicA" results)]. Ter Arkh. 2020 Oct 14;92(9):30-38. doi: 10.26442/00403660.2020.09.000699. Russian. PMID 33346428